CLINICAL TRIAL: NCT01553123
Title: A Randomized, Placebo Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Ulipristal Acetate in Women With Anemia Associated With Uterine Leiomyomas
Brief Title: Efficacy and Safety Study of Ulipristal Acetate in Females With Anemia Associated With Uterine Leiomyoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UL1104
Record Dates: First submitted 2012-03-02; First posted 2012-03-13 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Leiomyomas
Keywords: Leiomyomas
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate; Iron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ulipristal with iron (Experimental)
  Interventions: Drug: Ulipristal Acetate; Drug: Iron
- Placebo (Placebo Comparator): Placebo with iron
  Interventions: Drug: Iron

INTERVENTIONS:
Drug: Ulipristal Acetate — once daily, oral
  Other Names: UPA
  Arms: Ulipristal with iron
Drug: Iron — once daily, dried ferrous sulfate

SUMMARY:
The purpose of this study is to determine whether ulipristal acetate is effective in the treatment of females with anemia associated with uterine leiomyomas. The safety of this product will also be evaluated.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, multicenter study with parallel groups in order to evaluate the efficacy and safety of ulipristal acetate in female subjects with anemia associated with uterine leiomyomas. The objective of this study is to determine if daily ulipristal acetate with iron is more effective than iron alone.

ELIGIBILITY:
Inclusion Criteria:

* Is a pre-menopausal female, 18 - 50 years;
* Has documented leiomyoma(s);
* Has leiomyoma-related anemia;
* Has an endometrial biopsy within the screening period prior to the first dose of the test article which shows no endometrial hyperplasia;
* Is willing and able to provide written informed consent and authorization to disclose protected health information.

Exclusion Criteria:

* Has a history of uterine surgery that would interfere with the study;
* Has a condition requiring immediate or intermittent blood transfusions;
* Has a known coagulation disorder;
* Has a history of uterine, cervix, ovarian, or breast cancer;
* Has used a selective progesterone receptor modulator or a gonadotrophin releasing hormone agonist in previous 6 months;
* Has received blood transfusion within 8 weeks before the screening visit;
* Has abnormal liver functions;
* Is pregnant.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin levels (g/dL) | Day 1 of the first on-treatment menstrual cycle to the start, or scheduled start of menstrual cycle 3.
  Change from baseline in hemoglobin levels (g/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Zobrist, MS, PhD, Study Director — Watson Pharmaceuticals
Locations (47):
- United States (47):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Coastal Clinical Research, Inc, Mobile, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Benchmark Research, Sacramento, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - All Women's Healthcare of West Broward, Plantation, Florida
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Atlanta Women's Research Institute, Inc, Atlanta, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Fellows Research Alliance, Savannah, Georgia
  - Women's Health Practice, Champaign, Illinois
  - Advanced Gynecologic Surgery Institute, Naperville, Illinois
  - Center for Women's Research, Palos Heights, Illinois
  - South Bend Clinical, Granger, Indiana
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - Women Under Study, LLC, New Orleans, Louisiana
  - Hutzel Womens Health Specialists, Detroit, Michigan
  - Women's Clinic of Lincoln, P.C., Lincoln, Nebraska
  - Office of Annette Mayes, MD, PC, Las Vegas, Nevada
  - Office of Edmond Pack, MD, Las Vegas, Nevada
  - Office of R. Garn Mabey, Jr, Las Vegas, Nevada
  - Lawrence Obstetrics-Gynecology Clinical Research, Lawrenceville, New Jersey
  - Southwest Clinical Research, Albuquerque, New Mexico
  - New York Center for Women's Health Research, New York, New York
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - Physicians for Women of Greensboro, Greensboro, North Carolina
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Hawthorne Medical Research, Winston-Salem, North Carolina
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Advanced Clinical Concepts, West Reading, Pennsylvania
  - Southeast Regional Research Group, Aiken, South Carolina
  - South Carolina Clinical Research Center, LLC, Columbia, South Carolina
  - Discovery Clinical Trials - Genesis Health Central Women's Care, Dallas, Texas
  - Advances in Health Inc, Houston, Texas
  - Willowbend Health and Wellness Associates, Plano, Texas
  - Clinical Trials of Texas Incorporated Laboratory, San Antonio, Texas
  - Riverside Regional Medical Center, Newport News, Virginia